CLINICAL TRIAL: NCT02606695
Title: A Prospective Multicenter Study Evaluating the Clinical and Radiographic Outcomes of Thoracolumbar Spine Surgery When Comprehensive Sagittal Alignment Surgical Planning is Used
Brief Title: Comprehensive Spinal Alignment Planning Study
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.IGA1503
Record Dates: First submitted 2015-11-05; First posted 2015-11-17 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Spine Surgery
Keywords: Spine Surgery Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- NuvaMap and NuvaMap OR in Thoracolumbar Spinal Fusion
  Interventions: Device: NuvaMap O.R.; Device: NuvaMap

INTERVENTIONS:
Device: NuvaMap O.R. — Clinical imaging software used to assess intraoperative spinal alignment
Device: NuvaMap — Clinical imaging software used to assess spinal alignment

SUMMARY:
A comprehensive approach to the evaluation of alignment in spinal surgery patients - through preoperative planning, intraoperative assessment, and postoperative confirmation - has not been well-studied. This study aims to assess the value of such planning through clinical and radiographic outcomes.

DETAILED DESCRIPTION:
Preoperative planning using tools such as NuvaMapTM (NuVasive®, Inc., San Diego, CA) enable a surgeon to preoperatively evaluate these alignment parameters and simulate a patient-specific plan using a combination of procedures, techniques, and implants. Once in the operating room, realignment objectives can be verified from a lateral fluoroscopic image in real-time using NuvaMap O.R. (NuVasive, Inc.), a software application integrated with the NVM5® neuromonitoring platform (NuVasive, Inc.). This real-time verification allows for confirmation and subsequent changing of the plan as necessary. The objective of this study is to validate the utility and effectiveness of comprehensive surgical planning in restoring and preserving sagittal alignment through the collection of clinical and radiographic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who are at least 18 years of age;
2. Patients with planned thoracolumbar (any number of levels between T1 and the pelvis) spine fusion surgery and available preoperative standing lateral radiographs, inclusive of the femoral head axis;
3. Able to undergo surgery based on physical exam, medical history and surgeon judgment;
4. Patients who understand the conditions of enrollment and are willing to sign an informed consent to participate in the evaluation.

Exclusion Criteria:

1. Patient has a mental or physical condition that would limit the ability to comply with study requirements;
2. Patient is a prisoner;
3. Patient is participating in another clinical study that would confound study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 300 patients will be enrolled in this multicenter observational study. The following eligibility criteria are designed to identify existing clinic patients for whom study under this protocol are considered appropriate. All subjects must meet the inclusion/exclusion criteria below in order to be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the utility of alignment planning using surgical planning software | Postoperative (3 months)
  The incidence of a change in plan (pre- or intraoperative) based on alignment measurement feedback, and the consequential achievement of postoperative (at 3 months) alignment relative to planned goals.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Scripps Clinic Medical Group, La Jolla, California
  - Orthopaedic Specialty Institute (OSI), Orange, California
  - Neurosurgical Medical Clinic, Inc., San Diego, California
  - Spine Colorado, Durango, Colorado
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Augusta Orthopedic & Sports Medicine Specialists, Augusta, Georgia
  - Rezin Orthopedics and Sports Medicine, Morris, Illinois
  - Dupage Medical Group Spine Institute, Naperville, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - University Spine Center, Wayne, New Jersey
  - Jacobs Institute/UB Neurosurgery, Inc.,, Amherst, New York
  - Spine Center at Great Neck, Great Neck, New York
  - Carolina Neurosurgery & Spine Associates (CNSA), Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Carilion Clinic (Roanoke), Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.nuvasive.com